CLINICAL TRIAL: NCT03322462
Title: A Multicenter Screening Study With Flortaucipir F 18 in Patients With Early Symptomatic AD
Brief Title: Tau Screening Study in Patients With Early Symptomatic AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A23
Record Dates: First submitted 2017-10-16; First posted 2017-10-26 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flortaucipir PET Scan (Experimental)
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET Scan

INTERVENTIONS:
Drug: Flortaucipir F18 — 370 megabecquerel (MBq) IV single-dose
  Other Names: 18F-AV-1451; [F-18]T807
Procedure: Brain PET Scan — positron emission tomography (PET) scan of the brain

SUMMARY:
This protocol is designed to serve as a pre-screening study for subjects who are potentially eligible for Alzheimer's Disease (AD) therapeutic trials that require tau imaging for inclusion by means of a flortaucipir F18 Positron Emission Tomography (PET) scan.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 60 and 85 years of age at the time of consent
* Patients with gradual and progressive change in memory function for a period equal to or greater than six months
* Patients who have a Mini Mental State Examination (MMSE) score in the 20-27 range
* Patients who are willing to undergo a PET scan using flortaucipir F 18
* Patients who give informed consent or have a legally authorized representative (LAR) to consent for enrollment

Exclusion Criteria:

* Patients who lack adequate premorbid literacy, vision, or hearing to complete the required psychometric testing in the investigator's opinion
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity, or not using reliable contraception methods. Females of childbearing potential must not be pregnant (negative serum β-Human Chorionic Gonadotropin [HCG] at screening and negative urine β-HCG prior to flortaucipir F 18 injection) or breastfeeding at screening. Females should agree to avoid becoming pregnant by refraining from sexual activity or using reliable contraceptive methods for 24 hours following flortaucipir F 18 injection administration.
* Have significant neurological disease affecting the Central Nervous System (CNS) (other than AD) that may affect cognition or ability to complete the study, including but not limited to, other types of dementia, serious brain infections, Parkinson's disease, multiple concussions, or epilepsy or recurrent seizures (except febrile childhood seizures).
* Patients with any current primary psychiatric diagnosis other than AD if, in the opinion of the investigator, the disorder/symptom is likely to confound interpretation of drug effect, affect cognitive assessment, or affect the patient's ability to complete the study (patients with history of schizophrenia or other chronic psychosis are excluded).
* Intend to use drugs known to significantly prolong the QT interval within 14 days or 5 half-lives (whichever is longer) of a scheduled screening/baseline flortaucipir F 18 PET scan, or have medical history of risk factors for Torsades du Pointes.
* Have an average electrocardiography (ECG) corrected QT (QTcF) interval measurement > 450 msec (men) or > 470 msec (women) at screening (as determined at the investigational site).
* Have ocular pathology that significantly limits ability to reliably evaluate vision or the retina.
* Have a history of alcohol or drug disorder (except tobacco use disorder) within 2 years before the screening visit
* Have a current serious or unstable illness including retinal, cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic (other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses in this study; or has a life expectancy of less than 24 months.
* Has a history of cancer within the last five years, with the exception of non-metastatic basal and/or squamous cell carcinoma of the skin, in situ cervical cancer, non-progressive prostate cancer, or other cancers with low risk of recurrence or spread
* Patients with a past history (suspected or confirmed) of Hepatitis B or Hepatitis C
* History of vitiligo and/or current evidence of post-inflammatory hypopigmentation
* Have had prior treatment with a passive anti-amyloid immunotherapy less than five half-lives prior to randomization.
* Have previously participated in any other study investigating active immunization against amyloid beta (Aβ)
* Patients that are currently enrolled in any other interventional clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Contraindication to PET
* Has hypersensitivity to flortaucipir F 18 or any of its excipients
* Present or planned exposure to ionizing radiation that, in combination with the planned administration of study PET ligands, would result in a cumulative exposure that exceeds local recommended exposure limits
* Has previous magnetic resonance imaging (MRI) evidence of significant abnormality that would suggest another potential etiology for progressive dementia or a clinically significant finding that may impact patient's potential to safely participate in study
* Have contraindications for MRI, including claustrophobia or the presence of contraindicated metal (ferromagnetic) implants/cardiac pacemaker
* Have poor venous access
* Are investigator site personnel directly affiliated with this study and/or immediate families; immediate family is defined as a spouse, parent, child, or sibling (biological or legally adopted)
* Are Lilly employees or are employees of third-party organizations (TPOs) involved in a study that requires exclusion of their employees
* Are otherwise unsuitable for a study of this type in the opinion of the investigator
* Have received treatment with a stable dose of an acetylcholinesterase inhibitor (AChEI) and/or memantine for less than two months before randomization (if a patient has recently stopped an AChEI and/or memantine, he/she must have discontinued treatment at least two months before randomization).
* Current use of strong inducers of CYP3A
* Are currently on medication(s) known to significantly prolong the QT interval
* Have allergies to either monoclonal antibodies, diphenhydramine, epinephrine, or methylprednisolone
* Have known allergies to LY3002813, related compounds, or any components of the formulation; or history of significant atopy
* Have known allergies to LY3202626, related compounds, or any components of the formulation
* Changes in concomitant medications that could potentially affect cognition and their dosing should be stable for at least one month before screening, and between screening and randomization (does not apply to medications discontinued due to exclusions or with limited duration of use, such as antibiotics)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (10):
- United States (9):
  - Pacific Research Network, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Brain Matters Research, Delray Beach, Florida
  - Bioclinica (Compass Research), Orlando, Florida
  - Axiom Clinical Research, Tampa, Florida
  - Boston Center for Memory, Newton, Massachusetts
  - PMG Research, Winston-Salem, North Carolina
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - The Memory Clinic, Bennington, Vermont
- Toronto Memory Program, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between Nov 2017 and Aug 2018. Recruited subjects with clinically diagnosed early AD who were interested in participating in AD therapeutic clinical trial AACG (Eli Lilly and Company; TRAILBLAZER-ALZ; NCT03367403)
Groups:
- Early Symptomatic AD Subjects: Early Symptomatic AD subjects in the flortaucipir PET scan arm
Period: Overall Study
Arm/Group | Early Symptomatic AD Subjects
Started | 155
Flortaucipir PET Scan | 155
Completed | 152
Not Completed | 3
Not completed — Technical difficulties | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Early Symptomatic AD Subjects
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 137
  More than one race | 0
  Unknown or Not Reported | 0
MMSE [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 24.5 (2.18)

OUTCOME MEASURES:

1. Primary Outcome: Flortaucipir Qualitative Results (Visual Reads)
Description: Flortaucipir PET scans were rated visually by an expert reader as follows: Not consistent with an AD pattern (τAD-), Moderate AD pattern (τAD+), or Advanced AD pattern and likely to progress (τAD++). Eligibility for AACG study was determined from the flortaucipir PET scan quantitation (SUVr; see below) according to protocol-specified criteria that excluded subjects with tau PET signal that was above or below study criteria.
Time Frame: baseline scan
Population: Includes all subjects who completed the study with valid flortaucipir PET scan (n=152)
Measure: Count of Participants; unit: Participants
Groups:
- Early Symptomatic AD, Eligible for AACG Study: Subjects determined to be eligible for the AACG Study from the flortaucipir PET scan arm.
- Early Symptomatic AD, Ineligible for AACG Study: Subjects who were not eligible for the AACG Study from the flortaucipir PET scan arm.
- Early Symptomatic AD (Total): All subjects with early symptomatic AD from the flortaucipir PET scan arm
Arm/Group | Early Symptomatic AD, Eligible for AACG Study | Early Symptomatic AD, Ineligible for AACG Study | Early Symptomatic AD (Total)
Number analyzed (Participants) | 58 | 94 | 152
Participants
  τAD++, advanced AD pattern | 56 | 22 | 78
  τAD+, moderate AD pattern | 2 | 8 | 10
  τAD-, pattern not consistent with AD | 0 | 64 | 64

2. Primary Outcome: Flortaucipir Quantitative Results (SUVr)
Description: Flortaucipir standardized uptake value ratio (SUVr). A value of 1 signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain. Visual read categories as described for previous measure. Eligibility for AACG study was determined from the flortaucipir PET scan quantitation (SUVr; see below) according to protocol-specified criteria that excluded subjects with tau PET signal that was above or below study criteria.
Time Frame: baseline scan
Population: SUVr was not collected for patients with a τAD- result
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Arm/Group | Early Symptomatic AD, Eligible for AACG Study | Early Symptomatic AD, Ineligible for AACG Study | Early Symptomatic AD (Total)
Number analyzed (Participants) | 58 | 30 | 88
standardized uptake value ratio (SUVr)
  SUVr all | 1.21207 (0.119729) | 1.48576 (0.316435) | 1.30537 (0.244527)
  SUVr τAD++ subjects: number analyzed (Participants) | 56 | 22 | 78
  SUVr τAD++ subjects | 1.21518 (0.120696) | 1.65880 (0.143067) | 1.34031 (0.237395)
  SUVr τAD+ subjects: number analyzed (Participants) | 2 | 8 | 10
  SUVr τAD+ subjects | 1.12490 (0.012021) | 1.00991 (0.023239) | 1.03291 (0.052789)

ADVERSE EVENTS:
Time Frame: 48 hours after study drug administration
Description: Adverse events (AEs) were collected at scan visits, regardless of attribution to study drug. End of study for AE reporting was 48 hours after the last study drug administration. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to study drug.
Groups:
- Safety Analysis Population: All subjects with early symptomatic AD from the flortaucipir PET scan arm who received one dose of flortaucipir
Arm/Group | Safety Analysis Population
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155
Other Adverse Events (participants affected / at risk) | 2/155
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Population (N=155)
diarrhoea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03322462/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT03322462/SAP_001.pdf